CLINICAL TRIAL: NCT06407388
Title: Ultrasound Findings Predictive of Neonatal Outcomes in Diabetic Pregnancies
Brief Title: Ultrasound Findings in Diabetic Pregnancies
Status: Recruiting | Type: Observational
Sponsor: Eastern Virginia Medical School (Other)
Responsible Party: Principal Investigator, Alyssa Savelli-Binsted, Physician, Eastern Virginia Medical School
Other Study IDs: 23-03-FB-0061
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Criteria for inclusion of subjects
  * Patients who enter pregnancy with a diagnosis of type I or type II diabetes mellitus.
  * Pregnant women between the ages of 18-45
  * Live, singleton gestation
  * Understanding and ability to give informed consent
  Criteria for exclusion of subjects
  * Patient unwilling or unable to provide consent
  * Intrauterine fetal demise (no fetal heart beat identified and documented by two physicians)
  * Age less than 18 years of age
  * Multifetal gestation
  * Chromosomal abnormality
  * Congenital infection (Toxoplasmosis, Cytomegalovirus, Rubella, Varicella Zoster, Parvovirus B19
  * Major fetal congenital malformations (such as: major congenital heart defect, omphalocele, open neural tube defect, etc)
- Controls: The control group will be a referent population of the Human Placenta Project. This reference population consists of patients who meet the following criteria:
  Maternal:
  * Pregnancy Conceived Without Assisted Reproduction
  * Singleton gestation
  * Delivery: >37 0/7 weeks gestation
  * No gestational diabetes
  * No fetal growth restriction
  * No Smoking/ Alcohol/Drugs History;
  * Placenta Implantation: Normal
  * Fetal Umbilical Cord abnormalities: None;
  Fetal- Newborn Outcomes:
  * Gestational Age at Delivery: >37 0/7
  * No Congenital infection (Toxoplasmosis, Cytomegalovirus, Rubella, Varicella Zoster, Parvovirus B19
  * No Major fetal congenital malformations (such as: major congenital heart defect, omphalocele, open neural tube defect, etc)
  * Fetal -Newborn Weight >10 percentile ( no Hx of FGR or SGA)

SUMMARY:
The goal of our study is to identify ultrasonographic markers that can predict adverse neonatal outcomes. Specifically, we hypothesize that an increase in fetal liver volumes will increase transcutaneous bilirubin (TcB) in the newborn and thus jaundice requiring phototherapy. This information can be used in patient counseling and to guide future screening protocols for ultrasound in individuals with diabetes.

DETAILED DESCRIPTION:
This is a single center, prospective case control study. Cases will be collected prospectively and control subjects will be data collected retrospectively from the reference population of the human placenta project (IRB #15-09-FB-0179). If patients agree to participate, one ultrasound will be performed at 30-34 weeks' gestation to look at the fetal parameters as described below. It is standard of care for all patients with pregestational diabetes to receive growth ultrasounds throughout their pregnancy. Patients who are diagnosed with pregestational diabetes at EVMS routinely undergo an ultrasound at 30-34 weeks' gestation. Therefore, ultrasound data will be collected during their scheduled 30-34 week ultrasound visit and no additional ultrasounds will need to be performed. At the time of enrollment, the PI or other study collaborator will ensure that the patient has previously had a detailed ultrasound evaluation (Code 76811). These patients will then be followed prospectively until delivery. The neonates of the study patients will be followed via chart review after delivery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who enter pregnancy with a diagnosis of type I or type II diabetes mellitus.
* Pregnant women between the ages of 18-45
* Live, singleton gestation
* Understanding and ability to give informed consent

Exclusion Criteria:

* Patient unwilling or unable to provide consent
* Intrauterine fetal demise (no fetal heart beat identified and documented by two physicians)
* Age less than 18 years of age
* Multifetal gestation
* Chromosomal abnormality
* Congenital infection (Toxoplasmosis, Cytomegalovirus, Rubella, Varicella Zoster, Parvovirus B19
* Major fetal congenital malformations (such as: major congenital heart defect, omphalocele, open neural tube defect, etc)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: We plan to recruit 52 individuals with diabetes and 104 control subjects from the reference population of the human placenta project (IRB #15-09-FB-0179).
Sampling Method: Non-Probability Sample
Enrollment: 156 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Elevated TcB | June 2023 to June 2025
  The primary objective of this study is to identify if increased fetal liver volumes correlate with elevated transcutaneous bilirubin (TcB) in neonates of mothers with diabetes.

SECONDARY OUTCOMES:
Respiratory Distress | June 2023 to June 2025
  One or more signs of increased work of breathing, such as tachypnea with a respiratory rate > 60 breaths per minute, nasal flaring, chest retractions, or grunting [13] requiring oxygen support
Jaundice | June 2023 to June 2025
  Jaundice requiring phototherapy
Hypoglycemia | June 2023 to June 2025
  <40 mg/dl in the first 24 hours of life
Polycythemia | June 2023 to June 2025
  Hematocrit >65% or hemoglobin >22 mg/dl

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Division of Maternal-Fetal Medicine, Eastern Virginia Medical School, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided